CLINICAL TRIAL: NCT00758706
Title: A Double-blind, Randomised, Placebo-controlled, Parallel Group Multi-centre Phase IIa Study to Assess the Effects on Biomarkers in Induced Sputum, Bood and Uine of AZD1236 Administered as Oral Tablet in Moderate to Severe COPD Patients During a 6 Week Period.
Brief Title: A Phase IIa Study Assessing the Effects of AZD1236 on Biomarkers in Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: BICO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4260C00007
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 4-((5-chloro-2-pyridinyl)oxy)-1-((((4S)-4-methyl-2,5-dioxo-4-imidazolidinyl)methyl)sulfonyl)-piperidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1236 (Experimental): oral tablet, 75 mg, twice daily during 6 weeks
  Interventions: Drug: AZD1236
- Placebo (Placebo Comparator): Dosing to match AZD1236
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1236 — oral tablet, 75 mg, twice daily during 6 weeks
  Arms: AZD1236
Drug: Placebo — Dosing to match AZD1236
  Arms: Placebo

SUMMARY:
The primary aim of this study is to investigate the effects of AZD1236 compared with placebo ("inactive substance") in COPD patients by analysing biomarkers for inflammation and tissue degradation in blood, urine and sputum.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD for 1 month
* Men or postmenopausal women
* Spirometry values indicating symptomatic patients
* Smoking history equivalent to using 20 cigarettes a day for 10 years.

Exclusion Criteria:

* Any current respiratory tract disorders other than COPD
* Requirement for regular oxygen therapy
* Acute worsening of COPD (exacerbation) 1,5 month prior to study drug administration
* Use of oral or parenteral glucocorticosteroids within 30 days and use of inhaled steroids 14 days prior to the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Dahl, MD, Professor, Principal Investigator — Arhus Kommune HospitalMedicinsk; Andrew Lockton, MD, Study Director — AstraZeneca R&D Charnwood
Locations (10):
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Arhus C
  - Research Site, København NV
  - Research Site, Odense C
- Finland (2):
  - Research Site, Helsinki
  - Research Site, Tampere
- Netherlands (2):
  - Research Site, Eindhoven
  - Research Site, Nieuwegein
- Norway (2):
  - Research Site, Oslo
  - Research Site, Trondheim

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=360&filename=CSR-D4260C00007.pdf
- See also: D4260C00007 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=360&filename=CSR-D4260C00007.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD1236: AZD1236 75mg oral tablet twice daily(bid)
- Placebo: Placebo to AZD1236 twice daily(bid)
Period: Overall Study
Arm/Group | AZD1236 | Placebo
Started | 26 | 29
Completed | 22 | 25
Not Completed | 4 | 4
Not completed — Adverse Event | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1236 | Placebo | Total
Number analyzed (Participants) | 26 | 29 | 55
Age, Continuous [Mean (Full Range); unit: Year] | 62.9 [47 to 80] | 65.7 [49 to 79] | 64.1 [47 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Ratio of TNF Alpha at Week 6 to Baseline
Description: Ratio reflects Sputum Tumor Necrosis Factor alpha (TNF alpha) at week 6 value divide by baseline value. Baseline is geometric mean of Visit 2 (last value during run-in) and Visit 3 (Randomization).
Time Frame: Baseline and Week 6
Population: Full analysis set excluded participants without baseline or post-baseline data.
Measure: Mean (Full Range); unit: ratio
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 23 | 27
ratio | 1.37 (0.532) [0.532 to 18.7] | 1.21 (0.270) [0.270 to 20.4]

2. Primary Outcome: Ratio of Sputum Total Cells at Week 6 to Baseline
Description: Ratio reflects Sputum Total Cells at week 6 value divide by baseline value. Baseline is geometric mean of Visit 2 (last value during run-in) and Visit 3 (Randomization).
Time Frame: Baseline and Week 6
Population: Full analysis set excluded participants without baseline or post-baseline data.
Measure: Mean (Full Range); unit: ratio
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 23 | 27
ratio | 1.07 (0.209) [0.209 to 4.03] | 0.876 (0.002) [0.002 to 13.5]

3. Primary Outcome: Ratio of Total Urine Desmosine at Week 6 to Baseline
Description: Ratio reflects Total Urine Desmosine at week 6 value divide by baseline value. Baseline is visit 3(Randomization) value.
Time Frame: Baseline and Week 6
Population: Full analysis set excluded participants without baseline or post-baseline data.
Measure: Mean (Full Range); unit: ratio
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 24 | 28
ratio | 0.946 (0.240) [0.240 to 5.44] | 1.27 (0.387) [0.387 to 5.73]

4. Secondary Outcome: Incidence of Adverse Events
Description: Number of patients who had an AE
Time Frame: all study visits
Measure: Number; unit: Participants
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 26 | 29
Participants | 15 | 15

5. Secondary Outcome: Change From Baseline in Forced Expiratory Volume (FEV1) at Week 6
Description: Change from baseline reflects the Week 6 value minus the baseline value. Baseline is visit 3(randomization) value.
Time Frame: Baseline and Week 6
Population: Full analysis set completed at week 6
Measure: Mean (Full Range); unit: L
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 26 | 28
L | -0.025 (-0.510) [-0.510 to 0.670] | -0.063 (-0.670) [-0.670 to 0.550]

6. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Week 6
Description: Change from baseline reflects the Week 6 value minus the baseline value. Baseline is visit 3(randomization) value.
Time Frame: Baseline and Week 6
Population: Full analysis set completed at week 6
Measure: Mean (Full Range); unit: L
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 26 | 28
L | -0.103 (-0.960) [-0.960 to 0.740] | -0.104 (-0.900) [-0.900 to 1.23]

7. Secondary Outcome: Change From Baseline in Vital Capacity (VC) at Week 6
Description: Change from baseline reflects the Week 6 value minus the baseline value. Baseline is visit 3(randomization) value.
Time Frame: Baseline and Week 6
Population: Full analysis set completed at week 6
Measure: Mean (Full Range); unit: L
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 25 | 28
L | 0.098 (-0.680) [-0.680 to 2.72] | -0.110 (-0.840) [-0.840 to 0.590]

8. Secondary Outcome: Change From Baseline in Inspiratory Capacity (IC) at Week 6
Description: Change from baseline reflects the Week 6 value minus the baseline value. Baseline is visit 3(randomization) value.
Time Frame: Baseline and Week 6
Population: Full analysis set completed at week 6
Measure: Mean (Full Range); unit: L
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 25 | 28
L | -0.082 (-0.700) [-0.700 to 0.500] | -0.173 (-2.19) [-2.19 to 0.840]

9. Secondary Outcome: Change From Baseline in Forced Expiratory Flow (FEF) 25-75% at Week 6
Description: Change from baseline reflects the Week 6 value minus the baseline value. Baseline is visit 3(randomization) value.
Time Frame: Baseline and Week 6
Population: Full analysis set completed at week 6
Measure: Mean (Full Range); unit: L/s
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 26 | 28
L/s | -0.007 (-0.410) [-0.410 to 0.260] | -0.067 (-0.780) [-0.780 to 0.230]

10. Secondary Outcome: Change From Baseline in Peak Expiratory Flow (PEF) Morning at Average of Last 4 Week Treatment
Description: Change from baseline reflects the average of last 4 week on treatment (Week 1, Week 2, Week 4 and Week 6) minus the baseline value. Baseline is the mean of the last 10 days of data during run-in.
Time Frame: Baseline and last 4 week on treatment(Week 1, Week 2, Week 4 and Week 6)
Population: Full analysis set
Measure: Mean (Full Range); unit: L/min
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 26 | 29
L/min | -9.81 (-61.2) [-61.2 to 26.2] | -7.73 (-73.2) [-73.2 to 43.4]

11. Secondary Outcome: Change From Baseline in Peak Expiratory Flow (PEF) Evening at Average of Last 4 Week Treatment
Description: as for outcome 10
Time Frame: Baseline and last 4 week on treatment(Week 1, Week 2, Week 4 and Week 6)
Population: Full analysis set
Measure: Mean (Full Range); unit: L/min
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 26 | 29
L/min | -13.6 (-80.3) [-80.3 to 30.1] | -13.5 (-102) [-102 to 27.4]

12. Secondary Outcome: Change From Baseline in Clinical COPD Questionnaire(CCQ) Total
Description: Change from baseline reflects the Week 6 value minus the baseline value. Baseline is visit 3(randomization) value. The total scores vary between 0 (never/not limited at all) to 6 (almost all the time/totally limited)
Time Frame: Baseline and Week 6
Population: Full analysis set
Measure: Mean (Full Range); unit: Score on scale
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale | 0.011 (-0.800) [-0.800 to 1.40] | -0.241 (-1.74) [-1.74 to 1.20]

13. Secondary Outcome: Change From Baseline in COPD Symptoms, Breathlessness at Average of Last 4 Week Treatment
Description: Change from baseline reflects the average of last 4 week on treatment (Week 1, Week 2, Week 4 and Week 6) minus the baseline value. Baseline is the mean of the last 10 days of data during run-in. Score vary between 0 (None) to 4 (Severe).
Time Frame: Baseline and last 4 week on treatment(Week 1, Week 2, Week 4 and Week 6)
Population: Full analysis set
Measure: Mean (Full Range); unit: Score on scale
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 26 | 29
Score on scale | -0.191 (-1.51) [-1.51 to 1.00] | -0.338 (-1.74) [-1.74 to 1.42]

14. Secondary Outcome: Change From Baseline in COPD Symptoms, Chest Tightness at Average of Last 4 Week Treatment
Description: as for outcome 13
Time Frame: Baseline and last 4 week on treatment(Week 1, Week 2, Week 4 and Week 6)
Population: Full analysis set
Measure: Mean (Full Range); unit: Score on scale
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 26 | 29
Score on scale | -0.149 (-1.11) [-1.11 to 1.00] | -0.156 (-1.74) [-1.74 to 1.27]

15. Secondary Outcome: Change From Baseline in COPD Symptoms, Cough Score at Average of Last 4 Week Treatment
Description: Change from baseline reflects the average of last 4 week on treatment (Week 1, Week 2, Week 4 and Week 6) minus the baseline value. Baseline is the mean of the last 10 days of data during run-in. Score vary between 0 (None) to 4 (Almost Constant).
Time Frame: Baseline and last 4 week on treatment(Week 1, Week 2, Week 4 and Week 6)
Population: Full analysis set
Measure: Mean (Full Range); unit: Score on scale
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 26 | 29
Score on scale | -0.114 (-1.81) [-1.81 to 1.78] | -0.324 (-1.94) [-1.94 to 1.13]

16. Secondary Outcome: Change From Baseline in COPD Symptoms, Night Time Awakenings at Average of Last 4 Week Treatment
Description: as for outcome 15
Time Frame: Baseline and last 4 week on treatment(Week 1, Week 2, Week 4 and Week 6)
Population: Full analysis set
Measure: Mean (Full Range); unit: Score on scale
Arm/Group | AZD1236 | Placebo
Number analyzed (Participants) | 26 | 29
Score on scale | 0.072 (-0.556) [-0.556 to 1.38] | -0.150 (-2.22) [-2.22 to 0.976]

ADVERSE EVENTS:
Arm/Group | AZD1236 | Placebo
Serious Adverse Events (participants affected / at risk) | 4/26 | 0/29
Other Adverse Events (participants affected / at risk) | 7/26 | 10/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1236 (N=26) | Placebo (N=29)
Exacerbation COPD (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Increased Dyspnoe After Stopping Normal Treatment (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decompensation Cordis (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1236 (N=26) | Placebo (N=29)
COPD (Respiratory, thoracic and mediastinal disorders) | 3 | 3
influenza (Infections and infestations) | 1 | 3
nasopharyngitis (Infections and infestations) | 1 | 3
oedema peripheral (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less